CLINICAL TRIAL: NCT05814874
Title: Human Intervention Study on the Improvement of the Selenium Supply in a Vegan Diet by Different Selenium Sources
Brief Title: Improvement of the Selenium Supply in a Vegan Diet by Different Selenium Sources
Acronym: SelVeg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Anna Kipp, Prof. Dr., University of Jena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-2913-BO
Record Dates: First submitted 2023-03-23; First posted 2023-04-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-01

CONDITIONS: Diet, Vegan; Selenium
MeSH Terms: interventions — 2S albumin, brazil nut

STUDY DESIGN:
Intervention Model Description: non-blinded randomized controlled trial Parallel group design (2 groups): vegan (exclusion of animal products) vs. omnivore (weekly consumption of meat and/or sausage), stable dietary habit since at least one year, 3 intervention groups (placebo, Brazil nut or selenium supplement)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- meat-based diet; placebo (Placebo Comparator)
  Interventions: Other: Placebo
- meat-based diet; selenium supplement (Active Comparator)
  Interventions: Dietary Supplement: selenium supplement
- meat-based diet; Brazil nut (Active Comparator)
  Interventions: Dietary Supplement: Brazil nut
- vegan diet; placebo (Placebo Comparator)
  Interventions: Other: Placebo
- vegan diet; selenium supplement (Active Comparator)
  Interventions: Dietary Supplement: selenium supplement
- vegan diet; Brazil nut (Active Comparator)
  Interventions: Dietary Supplement: Brazil nut

INTERVENTIONS:
Dietary Supplement: selenium supplement — Selenium supplement containing 55 µg of sodium selenate
  Arms: meat-based diet; selenium supplement; vegan diet; selenium supplement
Dietary Supplement: Brazil nut — Brazil nut butter; consumption corresponds to a selenium intake of 55 µg/d
  Arms: meat-based diet; Brazil nut; vegan diet; Brazil nut
Other: Placebo — Placebo pill
  Arms: meat-based diet; placebo; vegan diet; placebo

SUMMARY:
As vegans are among the individuals with the lowest serum selenium levels, the randomized controlled SelVeg study aims to address the question of whether Brazil nuts could be an adequate source of selenium for diets potentially low in selenium. For this purpose, we will investigate in individuals with a vegan or omnivorous dietary pattern how a daily selenium intervention in the form of a food (here Brazil nut butter) or an over-the-counter selenium supplement affects the selenium status.

DETAILED DESCRIPTION:
The vegan diet is characterized by an exclusion of all animal foods and is associated with positive health effects. However, dietary restriction can lead to inadequate intake of both macro- and micronutrients. Selenium and zinc, among others are critical nutrients in a vegan diet. Brazil nuts represent a particularly selenium-rich plant food. In addition to selenium Brazil nuts have also relevant amounts of other trace elements, including zinc, iron and copper.

Therefore, the aim of this study is to evaluate the effect of a daily selenium supplementation in the form of Brazil nut butter in comparison to a selenium supplement. As primary outcome, the serum selenium concentration and other serum biomarkers of the selenium status will be analyzed. Additionally, serum levels of other trace elements such as zinc will be quantified. Dietary questionnaires will provide information on dietary intake of nutrients (focus on dietary fiber, zinc and phytate intake) to identify potential factors influencing selenium bioavailability.

The SelVeg study will enroll 90 healthy subjects with either a vegan (defined as exclusion of animal products) or omnivore (defined as weekly consumption of meat and/or sausage) dietary pattern. After categorizing in vegans or omnivores, participants are than randomized in one of the three intervention groups (placebo, Brazil nut or selenium supplement) and will receive 55 µg of additional daily selenium (as Brazil nut butter or tablet) or no additional selenium in case of placebo. The intervention period is 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy participant
* Adherence to one of following eating habit (vegan or omnivore) confirmed by food frequency protocol (5 d), lifestyle and nutrition questionnaires
* Stable eating habit for at least 1 year before enrollment

Exclusion Criteria:

* Diet other than omnivore or vegan
* Changing diet during the study period
* Baseline serum selenium concentration > 150 µg/L
* Acute or chronic disease (tumor, infection, other), gastrointestinal diseases, chronic renal disease, diseases of the parathyroids, diseases necessitating regular phlebotomies
* Nut allergy
* Pregnancy or lactation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female (before menopause) and male gender (50% each)
Enrollment: 90 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Selenium status | baseline and after 2 weeks
  Changes in serum selenium concentration [µg/L] and selenoprotein-based biomarkers (SELENOP and GPX [U/L]) after intervention

SECONDARY OUTCOMES:
Trace element serum concentrations | baseline and after 2 weeks
  Change in serum concentration of trace elements (zinc, copper, manganese, iron, potassium and calcium [µg/L]) after intervention
Anthropometric data | baseline and after 2 weeks
  body mass index [kg/m2]
Mean macro- and micronutrient intake over 5 days | baseline
Dietary zinc and phytate intake | 6 months
  Zinc and Phytate Diet Score (= frequency index * quantity index * zinc or phytate content [mg])

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich Schiller University Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Open access publications
Supporting Information: Study Protocol, SAP
Time Frame: end of 2023

REFERENCES:
- [Derived] Simon R, Lossow K, Pellowski D, Kipp K, Achatz M, Klasen N, Schwerdtle T, Dawczynski C, Kipp AP. Improving the selenium supply of vegans and omnivores with Brazil nut butter compared to a dietary supplement in a randomized controlled trial. Eur J Nutr. 2025 Feb 1;64(2):74. doi: 10.1007/s00394-025-03587-z. PMID 39891729